CLINICAL TRIAL: NCT06290141
Title: A Phase 3, Randomized, Double-blind, Study Evaluating Efficacy and Safety of Riliprubart Versus Intravenous Immunoglobulin (IVIg) in Participants With Chronic Inflammatory Demyelinating Polyneuropathy
Brief Title: A Study to Test the Efficacy and Safety of Riliprubart Against the Usual Treatment of Intravenous Immunoglobulin (IVIg) in People With Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Acronym: VITALIZE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC18156; U1111-1295-3363 (Registry Identifier: ICTRP); 2023-508338-33 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Intervention Model Description: Part A is a double-blind treatment period and Part B is an open-label period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Riliprubart Arm (Experimental): Riliprubart + Placebo IVIg for 24 weeks followed by open-label extension phase with riliprubart for 24 weeks
  Interventions: Drug: riliprubart; Drug: Placebo
- IVIg Arm (Active Comparator): IVIg (IVIg continuation) + Placebo riliprubart for 24 weeks followed by open-label extension phase with riliprubart for 24 weeks
  Interventions: Drug: Placebo; Drug: riliprubart; Drug: IVIg

INTERVENTIONS:
Drug: riliprubart — Pharmaceutical form: Solution Route of administration: IV solution
  Other Names: SAR445088
  Arms: Riliprubart Arm
Drug: Placebo — Pharmaceutical form: Solution Route of administration: IV solution
  Arms: IVIg Arm
Drug: riliprubart — Pharmaceutical form: Solution Route of administration: SC solution
  Other Names: SAR445088
Drug: Placebo — Pharmaceutical form: Solution Route of administration: SC solution
  Arms: IVIg Arm
Drug: IVIg — Pharmaceutical form: Concentrate for solution for infusion (or any other formulation approved locally) Route of administration: IV solution
  Arms: IVIg Arm
Drug: Placebo — Pharmaceutical form: Placebo to match intravenous immunoglobulin IVIg for IV infusio Route of administration: IV solution
  Arms: Riliprubart Arm

SUMMARY:
The purpose of the study is to evaluate efficacy of riliprubart compared to IVIg in adult participants with CIDP who are receiving maintenance treatment with IVIg. The study duration will be for a maximum of 109 weeks including screening, treatment phases, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Participant must have CIDP or possible CIDP criteria, based on European Academy of Neurology (EAN)/ Peripherial Nerve Society (PNS) Task Force CIDP guidelines, second revision (2021).
2. Participant must have either typical CIDP, or one of the following 2 CIDP variants: motor CIDP (including motor-predominant CIDP), multifocal CIDP (also known as Lewis Sumner Syndrome). Diagnosis must be confirmed by the study adjudication committee.
3. Participants must have responded to IVIg in the past 5 years. Response must be an objective clinically meaningful improvement defined by at least one of the following: ≥1 point decrease in adjusted INCAT score, ≥4 points increase in I-RODS centile score, ≥3 points increase in the MRC-SS, ≥8 kilopascal improvement in mean grip strength (1 hand), or an equivalent improvement based on information documented in medical records as per the Investigator's judgment.
4. Participant must be on a stable maintenance dosage of IVIg, defined as no change greater than 10% in frequency or dose of IVIg within 8 weeks prior to Screening, and remaining stable until baseline.
5. Participant must have residual disability, defined as an INCAT score of 2 to 9 at Screening that is confirmed at baseline (a score of 2 should be exclusively from leg disability component of INCAT).
6. Participant must be receiving treatment with IVIg within a standard maintenance dosing regimen, defined as per EAN/PNS 2021 CIDP guidelines: 0.4 to 1 g/kg every 2 to 6 weeks. The IVIg maintenance dosing regimen should be equivalent or higher than a weekly dose of 0.1 g/kg body weight (for example, 0.3 g/kg every 3 weeks).
7. Participants receiving IVIg infusions at home are eligible, as long as IVIg infusions are switched to a hospital or infusion center setting at least 1 cycle prior to baseline.
8. Participant must have active disease, defined by a CIDP disease activity score (CDAS) of ≥2 points at Screening.
9. Participant must have documented vaccinations against encapsulated bacterial pathogens given within 5 years prior to Day 1 or initiated a minimum of 14 days prior to first dose of study intervention.
10. All participants must agree to use contraception methods during and after the study as required.
11. Contraceptive use by men and women participating in the study should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
12. A male participant is eligible to participate if they agree to the following during the study intervention period and for at least 55 weeks after the last dose of study medication.

    --Refrain from donating or cryopreserving sperm.

    PLUS, either:

    --Be abstinent from heterosexual intercourse (abstinent on a long-term and persistent basis) and agree to remain abstinent.

    OR

    --Must agree to use contraception/barrier as detailed below:
13. A male condom and an additional highly effective contraceptive method (Contraceptive and barrier guidance per protocol) when having sexual intercourse with a woman of childbearing potential (WOCBP) who is not currently pregnant.
14. A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies:

    * Is a woman of nonchildbearing potential (WONCBP) as defined by the protocol. OR
    * Is a WOCBP and agrees to use a contraceptive method that is highly effective (with a failure rate of <1% per year), as described in the protocol during the study intervention period (to be effective before starting the intervention) and for at least 55 weeks after the last administration of study intervention and agrees not to donate or cryopreserve eggs (ova, oocytes) for the purpose of reproduction during this period.
15. Participant must have a body weight at Screening of 35 kg to 154 kg (77 to 340 lbs) inclusive.
16. Evidence of at least one clinically meaningful deterioration within 2 years, or at least 2 clinically meaningful deteriorations within 5 years prior to screening which occurred during period of interrupted dosing, reduced dosage, or extended intervals between doses of immunoglobin therapy, as verified by clinical examination or medical records.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Polyneuropathy of other causes, including but not limited to acute demyelinating polyneuropathies (eg. Guillain-Barré syndrome), hereditary demyelinating neuropathies, neuropathies secondary to infection or systemic disease, diabetic neuropathy, drug- or toxin-induced neuropathies, multifocal motor neuropathy, polyneuropathy related to IgM monoclonal gammopathy, POEMS syndrome, lumbosacral radiculoplexus neuropathy.
2. Sensory CIDP, distal CIDP and focal CIDP variants.
3. Any other neurological or systemic disease that can cause symptoms and signs interfering with treatment or outcome assessments.
4. Poorly controlled diabetes (HbA1c glycated hemoglobin >7% at the Screening visit).
5. Serious infections requiring hospitalization within 30 days prior to Screening, any active infection requiring treatment during Screening, or presence of a condition that may predispose the participant to increased risk of infection (eg, medical history such as known immunodeficiency or history of recurrent infections).
6. Clinical diagnosis of Systemic Lupus Erythematosus (SLE) or family history of SLE. For a participant with an antinuclear antibody (ANA) titer ≥1:160 and a positive anti double-stranded DNA (anti-dsDNA) at Screening, SLE diagnosis must be ruled out prior to enrollment.
7. Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study. Specifically, history of any hypersensitivity reaction to riliprubart or its components or of a severe allergic or anaphylactic reaction to any humanized or murine monoclonal antibody.
8. Any contraindication related to the administration of immunoglobulins (eg hypersensitivity, chronic kidney disease, thromboembolic diseases or recent thromboembolic event, known history of IgA deficiency at the time of Screening).
9. Any other clinically meaningful medical history or ongoing medical condition (as determined by the Investigator at Screening) that might impact the benefit-risk assessment, jeopardize the safety of the participant, or compromise the quality of the data collected in this study; or history or presence of other significant concomitant illness that would adversely affect participation in this study, per the Investigator's judgment.
10. Documented history of attempted suicide over the 6 months prior to the Screening visit, presence of suicidal ideation of category 4 or 5 on the C-SSRS during Screening, OR if in the Investigator's judgment, the participant is at risk for a suicide attempt.
11. Evidence of CIDP worsening within the 6 weeks following a prior vaccination that, in the opinion of the Investigator, constituted a relapse.
12. Recent or planned major surgery that could confound the results of the trial or put the participant at undue risk.
13. Treatment with plasma exchange within 8 weeks prior to Screening.
14. Treatment within 3 months prior to dosing with immunosuppressive/ immunomodulator medication, or corticosteroids (except ≤20 mg/day of prednisone or equivalent which is allowed), or prior treatment (at any time) with highly immunosuppressive/ chemotherapeutic medications with sustained effects (eg, mitoxantrone, alemtuzumab, or cladribine).
15. Prior treatment with riliprubart.
16. Use of any specific complement system inhibitor (eg, eculizumab) within 12 weeks or 5 times the half-life of the product, whichever is longer, prior to Screening.
17. Prior treatment (any time) with total lymphoid irradiation or bone marrow transplantation.
18. Prior treatment with B-cell depleting agents such as rituximab within 6 months prior to riliprubart dosing, or until return of B-cell counts to normal levels, whichever is longer.
19. Any vaccination received within 28 days prior to dosing (with few exceptions to be confirmed at screening).
20. Participation in another clinical trial with an investigational drug or receipt of an investigational product within 12 weeks or 5 times the half-life of the product (whichever is longer) prior to Screening.
21. Any Screening laboratory values outside normal limits or abnormal ECG considered in the Investigator's judgment to be clinically significant in the context of this trial.
22. Positive result of any of the following tests:

    * HBsAg
    * Anti-HBc; unless anti-HBs Ab X are also positive, indicating natural immunity.
    * Anti-HCV antibodies.
    * Anti-HIV1 and anti-HIV2 antibodies.
23. Pregnancy, defined as a positive result of a highly sensitive urine or serum pregnancy test, or lactation.
24. Accommodation in an institution because of regulatory or legal order; imprisoned or legally institutionalized.
25. Participant not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures.
26. Participants are employees of the clinical study site or other individuals directly involved in the conduct of the study, or immediate family members of such individuals.
27. Any country-related specific regulation that would prevent the participant from entering the study as defined by the protocol.
28. Treatment with efgartigimod within 8 weeks prior to screening.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2027-07-09 (Estimated); Study Completion 2029-01-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants experiencing a response | Baseline to week 24
  A response is defined as decrease of ≥1 point from baseline in adjusted INCAT disability score at Week 24
Percentage of participants randomized to riliprubart who responded during part A and had a lasting response during the open-label treatment extension period | Baseline to week 48
  Lasting response is defined as a decrease of ≥1 point in adjusted INCAT disability score

SECONDARY OUTCOMES:
Change from baseline in Rasch-built Overall Disability Scale (I-RODS) score | Baseline to week 24
Change from baseline in adjusted inflammatory neuropathy cause and treatment (INCAT) disability score | Baseline to week 24
Change from baseline in grip strength (kilopascals, dominant hand) | Baseline to week 24
Change from baseline in Medical Research Council Sum Score (MRC-SS) | Baseline to week 24
Change from baseline in the Rasch-built modified fatigue severity scale (RT-FSS) | Baseline to week 24
Percentage of participants experiencing a relapse | Baseline to week 24
  A relapse is defined as increase of ≥1 point from baseline in adjusted INCAT disability score
Change from baseline in the EuroQol 5 Dimension, 5-Level Health Scale (EQ-5D-5L) | Baseline to week 24
Number of participants with TEAEs, including SAEs and AESIs for Part A | Baseline to week 24
Number of participants with treatment-emergent ADA in participants treated with riliprubart | Baseline to week 24
Number of participants with TEAEs, including SAEs and AESIs | Week 24 to week 48
Incidence and titer of anti-drug antibodies (ADA) during open-label treatment and follow-up | Baseline to week 109
Change from baseline in I-RODS | Baseline to week 48
Change from baseline in adjusted INCAT score | Baseline to week 48
Change from baseline in grip strength (kilopascals; dominant hand) | Baseline to week 48
Change from baseline in MRC-SS | Baseline to week 48
Change from baseline in EQ-5D-5L score | Baseline to week 48
Percentage of participants randomized to IVIg continuation who experienced a response | Week 24 to week 48
  A response is defined as a decrease of ≥1 point in adjusted INCAT disability scale score at Week 48 versus Week 24
Percentage of participants randomized to riliprubart who experienced a response at Week 48 without prior response in Part A (delayed response) | Baseline to Week 48
  A delayed response is defined as an decrease of ≥1 point in adjusted INCAT disability score at Week 48 versus Baseline
Percentage of participants randomized to riliprubart experiencing a relapse | Baseline to week 48
  A relapse is defined as an increase of ≥1 point from baseline in adjusted INCAT disability score at Week 48 versus Baseline
Change from baseline in RT-FSS | Baseline to week 48
Percentage of participants randomized to riliprubart experiencing a relapse | Week 24 to week 48
  A relapse is defined as a increase of ≥1 point from baseline in adjusted INCAT disability score at Week 48 versus Week 24.

CONTACTS AND LOCATIONS:
Locations (108):
- United States (23):
  - Alabama Neurology Associates- Site Number : 8400019, Homewood, Alabama
  - Honor Health Scottsdale Osborn Medical Center- Site Number : 8400014, Scottsdale, Arizona
  - Keck School of Medicine of University of Southern California- Site Number : 8400002, Los Angeles, California
  - University of California Irvine Medical Center- Site Number : 8400007, Orange, California
  - Yale University School of Medicine- Site Number : 8400018, New Haven, Connecticut
  - AdventHealth Orlando- Site Number : 8400006, Orlando, Florida
  - AdventHealth Site Number : 8400006, Orlando, Florida
  - NorthShore University Health System - Glenbrook Hospital- Site Number : 8400024, Glenview, Illinois
  - University of Kansas Medical Center- Site Number : 8400010, Kansas City, Kansas
  - Ochsner Medical Center - Jefferson Highway- Site Number : 8400030, New Orleans, Louisiana
  - Johns Hopkins Hospital- Site Number : 8400015, Baltimore, Maryland
  - Henry Ford Hospital- Site Number : 8400025, Detroit, Michigan
  - Michigan State University- Site Number : 8400038, East Lansing, Michigan
  - Washington University School of Medicine - Siteman Cancer Center- Site Number : 8400037, St Louis, Missouri
  - Dent Neurologic Institute - Amherst- Site Number : 8400039, Amherst, New York
  - Hospital for Special Surgery- Site Number : 8400041, New York, New York
  - Columbia University Irving Medical Center- Site Number : 8400003, New York, New York
  - University of Cincinnati Medical Center- Site Number : 8400020, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center- Site Number : 8400033, Cleveland, Ohio
  - Penn Medicine: University of Pennsylvania Health System- Site Number : 8400022, Philadelphia, Pennsylvania
  - Austin Neuromuscular Center- Site Number : 8400040, Austin, Texas
  - University of Vermont Medical Center- Site Number : 8400012, Burlington, Vermont
  - University of Virginia- Site Number : 8400023, Charlottesville, Virginia
- Argentina (3):
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320002, Buenos Aires
  - Investigational Site Number : 0320003, Buenos Aires
- Belgium (2):
  - Investigational Site Number : 0560002, Ghent
  - Investigational Site Number : 0560001, Leuven
- Brazil (4):
  - L2IP - Instituto de Pesquisas Clínicas- Site Number : 0760006, Brasília, Federal District
  - Instituto de Neurologia de Curitiba - Ecoville- Site Number : 0760007, Curitiba, Paraná
  - InsCer - Instituto do Cérebro da PUCRS- Site Number : 0760002, Porto Alegre, Rio Grande do Sul
  - PSEG Centro de Pesquisa Clínica- Site Number : 0760009, São Paulo
- Canada (3):
  - Investigational Site Number : 1240003, London, Ontario
  - Investigational Site Number : 1240006, Montreal, Quebec
  - Investigational Site Number : 1240001, Québec, Quebec
- China (17):
  - Investigational Site Number : 1560013, Beijing
  - Investigational Site Number : 1560010, Beijing
  - Investigational Site Number : 1560005, Beijing
  - Investigational Site Number : 1560017, Beijing
  - Investigational Site Number : 1560009, Changsha
  - Investigational Site Number : 1560011, Chengdu
  - Investigational Site Number : 1560002, Fuzhou
  - Investigational Site Number : 1560012, Guangzhou
  - Investigational Site Number : 1560007, Guangzhou
  - Investigational Site Number : 1560014, Hangzhou
  - Investigational Site Number : 1560016, Jiazhuang
  - Investigational Site Number : 1560008, Jinan
  - Investigational Site Number : 1560015, Nanchang
  - Investigational Site Number : 1560001, Shanghai
  - Investigational Site Number : 1560003, Wuhan
  - Investigational Site Number : 1560006, Wuhan
  - Investigational Site Number : 1560004, Xi'an
- Czechia (5):
  - Investigational Site Number : 2030004, Brno
  - Investigational Site Number : 2030003, Hradec Králové
  - Investigational Site Number : 2030005, Ostrava
  - Investigational Site Number : 2030002, Pardubice
  - Investigational Site Number : 2030001, Prague
- Denmark (2):
  - Investigational Site Number : 2080002, Aarhus
  - Investigational Site Number : 2080001, Copenhagen
- France (4):
  - Investigational Site Number : 2500001, Le Kremlin-Bicêtre
  - Investigational Site Number : 2500002, Marseille
  - Investigational Site Number : 2500005, Nice
  - Investigational Site Number : 2500003, Paris
- Germany (5):
  - Massachusetts General Hospital- Site Number : 8400009, Berlin, Massachusetts
  - Investigational Site Number : 2760003, Berlin
  - Investigational Site Number : 2760006, Göttingen
  - Investigational Site Number : 2760005, Hanover
  - Investigational Site Number : 2760001, Münster
- Hungary (3):
  - Investigational Site Number : 3480003, Budapest
  - Investigational Site Number : 3480004, Győr
  - Investigational Site Number : 3480001, Szeged
- Investigational Site Number : 3760001, Haifa, Israel
- Japan (9):
  - Investigational Site Number : 3920007, Amagasaki, Hyōgo
  - Investigational Site Number : 3920015, Yokohama, Kanagawa
  - Investigational Site Number : 3920012, Higashi-Matsuyama, Saitama
  - Investigational Site Number : 3920005, Kawagoe, Saitama
  - Investigational Site Number : 3920014, Yaizu, Shizuoka
  - Investigational Site Number : 3920008, Kodaira, Tokyo
  - Investigational Site Number : 3920010, Ōta-ku, Tokyo
  - Investigational Site Number : 3920001, Chiba
  - Investigational Site Number : 3920009, Saga
- Mexico (2):
  - Investigational Site Number : 4840002, Chihuahua City
  - Investigational Site Number : 4840001, Tlalnepantla
- Portugal (4):
  - Investigational Site Number : 6200003, Braga
  - Investigational Site Number : 6200005, Coimbra
  - Investigational Site Number : 6200002, Lisbon
  - Investigational Site Number : 6200001, Lisbon
- Spain (8):
  - Investigational Site Number : 7240009, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240006, Sabadell, Barcelona [Barcelona]
  - Investigational Site Number : 7240001, Barcelona, Catalunya [Cataluña]
  - Investigational Site Number : 7240008, Majadahonda, Madrid
  - Investigational Site Number : 7240002, Pamplona, Navarre
  - Investigational Site Number : 7240003, Oviedo, Principality of Asturias
  - Investigational Site Number : 7240007, Málaga
  - Investigational Site Number : 7240004, Valencia
- Investigational Site Number : 7520001, Stockholm, Sweden
- Switzerland (2):
  - Investigational Site Number : 7560001, Basel
  - Investigational Site Number : 7560003, Bern
- Taiwan (3):
  - Investigational Site Number : 1580003, Kaohsiung City
  - Investigational Site Number : 1580001, Taipei
  - Investigational Site Number : 1580002, Taipei
- Turkey (Türkiye) (4):
  - Investigational Site Number : 7920004, Bursa
  - Investigational Site Number : 7920001, Istanbul
  - Investigational Site Number : 7920002, Istanbul
  - Investigational Site Number : 7920003, Konya
- United Kingdom (3):
  - Investigational Site Number : 8260007, London, England
  - Investigational Site Number : 8260003, Inverness, Highland
  - Investigational Site Number : 8260001, Oxford, Oxfordshire

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC18156 (Vitalize) & EFC17236 (MOBILIZE) CIDP website-for potential participants — http://www.sanofistudies.com/G4SB
- See also: EFC18156 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25646&tenant=MT_SNY_9011